CLINICAL TRIAL: NCT06186440
Title: Cisplatin Plus Temozolomide Compared With Temozolomide in Patients With Newly Diagnosed MGMT Promotor Unmethylated Glioblastoma
Brief Title: Cisplatin Plus Temozolomide Compared With Temozolomide in Patients With MGMT Promotor Unmethylated Glioblastoma
Acronym: Glioblastoma
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Zhongnan Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: G32540
Record Dates: First submitted 2023-12-15; First posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Glioblastoma Multiforme of Brain
Keywords: Glioblastoma MGMT promoter unmethylation
MeSH Terms: interventions — Cisplatin; Temozolomide

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Cisplatin 20mg/m2 Cisplatin days 1-5 plus Temozolomide 150-200mg/m2 days 1-5
  Interventions: Drug: Cisplatin Plus Temozolomide
- Temozolomide (Active Comparator): Temozolomide 150-200mg/m2 days 1-5
  Interventions: Drug: Temozolomide

INTERVENTIONS:
Drug: Cisplatin Plus Temozolomide — Cisplatin Plus Temozolomide . Cisplatin 20mg/mCisplatin days 1-5
  Arms: Experimental
Drug: Temozolomide — Temozolomide
  Arms: Temozolomide

SUMMARY:
Temozolomide provided significant and clinically meaningful benefit in MGMT gene promoter methylation glioblastoma. However, in unmethylated patients, the effect of Temozolomide is limited. The aim of this study is to compare the effect of Cisplatin plus Temozolomide and Temozolomide in patients with MGMT gene promoter unmethylation glioblastoma

DETAILED DESCRIPTION:
60 Patients with glioblastoma were recruited for this study based on the following eligibility criteria: Age between 18 and 70, performance status of 0-1 (Eastern Cooperative Oncology Group performance status), histologically confirmed MGMT gene promoter unmethylation glioblastoma, no cerebrospinal fluid and distant metastatic disease. All patients had adequate hematologic, hepatic, and renal function. Patients younger than 18 years; patients with a prior (i.e. within 5 years) or synchronous malignancy, other than non-melanoma skin cancer; and those with significant comorbidities were excluded.

60 patients were randomly divided into two groups and compared the difference of efficacy between the two groups

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75, performance status of 0-1 (Eastern Cooperative Oncology Group performance status), histologically confirmed MGMT gene promoter unmethylation glioblastoma no cerebrospinal fluid and distant metastatic disease. adequate hematologic, hepatic, and renal function

Exclusion Criteria:

* younger than 18 years; with a prior (i.e. within 5 years) or synchronous malignancy, other than non-melanoma skin cancer; and those with significant comorbidities

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Estimated); Primary Completion 2024-12-01 (Estimated); Study Completion 2025-01-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 1 YEAR
  The length of time from the date of diagnosis to death from cancer

SECONDARY OUTCOMES:
PFS | 6 months
  the length of time after primary treatment for glioblastoma ends that the patient survives without any progression of glioblastoma

IPD SHARING:
Plan to Share IPD: No